CLINICAL TRIAL: NCT07318870
Title: Efficacy of Probenecid on Cluster Seizures During Anti Seizure Medication Withdrawal in Presurgical Focal Epilepsy Video-EEG Monitoring
Acronym: PROBCLUSTER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GHD_2024_12
Record Dates: First submitted 2025-12-04; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial | interventions — Probenecid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- probenecid (Experimental): Oral administration of PBN at a dose of 3g in adults or children weighting > 50 kg; at a dose of 2g in children weighting 35 to 50 kg; and at a dose of 1g in children weighting 20 to 34 kg.
  Interventions: Drug: Probenecid
- placebo (Placebo Comparator): Placebo administration in a scheme similar to experimental treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Probenecid — Oral administration of PBN at a dose of 3g in adults or children weighting > 50 kg; at a dose of 2g in children weighting 35 to 50 kg; and at a dose of 1g in children weighting 20 to 34 kg.
  Arms: probenecid
Other: Placebo — Placebo administration in a scheme similar to experimental treatment
  Arms: placebo

SUMMARY:
ProbCluster trial aims at making the proof of concept of antiseizure efficacy of the old antigout PBN in SC, in which Panx1 involvement is relevant on SC pathophysiology and in which efficient therapies are still lacking. The trial will be performed on patients with focal epilepsy in presurgical evaluation undergoing video-EEG monitoring, a setting characterized by a high risk of SC and an efficient video-EEG monitoring of seizures, reducing the risk of erroneous report based on patient home assessment. PBN is a good candidate for a repurposing in epilepsy, due to its brain penetration allowing Panx1 in situ blockade and of its good security profile. The repurposing process allows a faster, safer and cheaper development.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 6 and 50 years old
* weighting > 20 kg
* With focal seizures epilepsy
* Requiring video-EEG recording in Epilepsy Monitoring Units (EMU) for the presurgical evaluation of a focal epilepsy, with planned ASM withdrawal in order to precipitate seizure occurrence
* Able to take an oral therapy
* Ability to record the patient > 12 hours after the second seizure of the cluster
* Having received informed information about the study and having signed a consent form to participate in the study. Written consent of both holders of parental authority for minor patients.

Exclusion Criteria:

* Hypersensitivity to PBN or to any of the excipients (Microcrystalline cellulose, Hypromellose, Sodium carboxymethylamidon, Colloidal anhydrous silica, Magnesium stearate)
* Impaired renal function (creatinine clearance < 50 mL/min)
* Lithiasis diathesis
* Treatment by the following drugs: penicillins cephalosporins, acetylsalicylic acid, methotrexate, acetaminophen, naproxen, indomethacin, ketoprofen, meclofenamate, lorazepam, rifampicin, acyclovir, ganciclovir and zidovudine, sulfonamide, dyprophylline
* Acute gout attack
* Hyperuricemia secondary to cancer chemotherapy, radiotherapy or myeloproliferative neoplasia
* Primary hyperuricemia due to overproduction of uric acid.
* Pregnant or breast-feeding woman
* Patient benefiting from legal protection

Secondary exclusion criteria (before randomization) :

- Patient not randomized: Not experiencing at least 2 seizures lasting less than 10 minutes in 6 hours or less period (defining a SC) during the video-EEG monitoring period OR having no seizure recorded before the cluster.

Patients secondarily excluded will be excluded before randomization and will be replaced.

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Cessation of seizure recurrence in patients experiencing a cluster seizure | Time period from Day 0 to maximum Day 21
  Patients without seizure between 60 min and 12h after experimental treatment administration, assessed by the neurologist on video-EEG recording